CLINICAL TRIAL: NCT04375813
Title: Phase II Trial of Encapsulated Rapamycin (eRapa) for Bladder Cancer Prevention
Brief Title: Trial of Encapsulated Rapamycin (eRapa) for Bladder Cancer Prevention
Acronym: eRapa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Svatek (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Svatek, Professor, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00001422; R01CA252057 (NIH)
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multi-site phase II double-blind randomized trial. Subjects will be randomized into placebo arm or intervention arm with low dose (0.5 mg) eRapa (encapsulated rapamycin) Monday-Friday for one year or until disease recurrence. Patients will undergo endoscopic evaluation of the bladder every 3 months for 2 years, then every 6 months for 2 years, and at year 5. Some patients may also concurrently receive BCG immune therapy maintenance (weekly for 6 weeks for induction period, weekly for 3 weeks at 3 months, 6 months, and then every 6 months for a total of 7 maintenance cycles following tumor removal) per standard of care. Patient-reported outcome assessments, cognitive assessments, and physical assessments will be completed according to the study calendar. Research blood to assess safety, immune response and rapamycin level will be collected regularly throughout the study period. Participants will be followed for up to 5 years following enrollment.
Who Masked: Participant, Investigator
Masking Description: Once the list is generated, a non-study staff member will deliver the list to the designated pharmacist. The pharmacist will follow the generated list in consecutive order of enrollment to determine which group the subject will be assigned. The pharmacist will prepare the correct study drug (Placebo or eRapa (encapsulated rapamycin) 0.5 mg) and label the drug with subject information. Research staff will transport drug from pharmacy to clinic and provide for subject. Randomization will remain double blinded for study staff and subject. Patients will be given a once-daily oral eRapa (encapsulated rapamycin) at 0.5 mg or placebo MF for 1 year. Once the primary objectives have been met (i.e., all participants have completed follow up), the study staff and PI will be unblinded to the randomized study treatment arms. The above mentioned generated randomization list with subject assignments will be provided to the study staff and PI by the designated pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Study Drug Group (Active Comparator): Patients will be given 0.5mg eRapa (encapuslated rapamycin) orally each weekday (Monday-Friday) for one year.
  Interventions: Drug: eRapa
- Placebo Group (Placebo Comparator): Patients will be given a placebo (visually identical to the eRapa (encapsulated rapamycin)) orally each weekday (Monday-Friday) for one year.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: eRapa — 0.5mg eRapa (encapsulated rapamycin) oral capsules
  Other Names: encapsulated rapamycin
  Arms: Active Study Drug Group
Drug: Placebos — placebo capsules visually identical to eRapa oral capsules
  Arms: Placebo Group

SUMMARY:
eRapa (encapsulated rapamycin) will be investigated for secondary prevention in patients with diagnosed non-muscle invasive bladder cancer (NMIBC) through a phase II double-blind randomized controlled trial of long-term (one year) prevention with eRapa versus placebo. The primary hypothesis is that eRapa decreases the risk of cancer relapse for patients with NMIBC. Secondary hypotheses are that eRapa can improve certain immune parameters and improve cognition and physical function without adversely affecting patient-reported outcomes and quality of life.

DETAILED DESCRIPTION:
The study is a multi-site phase II double-blind randomized trial. Subjects will be randomized into placebo arm or intervention arm with low dose (0.5 mg) eRapa (encapsulated rapamycin) Monday-Friday for one year or until disease recurrence. Patients will undergo endoscopic evaluation of the bladder every 3 months for 2 years, then every 6 months for 2 years, and at year 5. Some patients may also concurrently receive BCG immune therapy maintenance (weekly for 6 weeks for induction period, weekly for 3 weeks at 3 months, 6 months, and then every 6 months for a total of 7 maintenance cycles following tumor removal) per standard of care. Patient-reported outcome (PRO) assessments, cognitive assessments, and physical assessments will be completed according to the study calendar. Research blood to assess safety, immune response and rapamycin level will be collected regularly throughout the study period. Participants will be followed for up to 5 years following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of non-muscle invasive (Ta, Tis, or T1) bladder cancer within 90 days prior to enrollment
* Able to give informed consent
* 18 years or older
* Patients must not be taking oral glucocorticoids at the time of registration
* Not have active, uncontrolled infections
* No other prior non-bladder malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.
* Patients with localized prostate cancer who are being followed by an active survelillance program are also eligible.
* Patients must not be pregnant or nursing, as the use of Intravesical BCG is not recommended during pregnancy. Women/ men of reproductive potential must have agreed to use an effective contraceptive method. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. Examples of effective contraception include hormonal contraception, double barrier method (condom with spermicidal cream, diaphragms with spermicidal cream, or condoms with diaphragms), Intrauterine device, and/or partner vasectomy. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. Both male and female patients will be required to disclose contraception method during screening and agree to continue to use that contraception method through the end of their participation in the study.
* Patients must have had all grossly visible papillary tumors removed within 90 days prior to registration or cystoscopy confirming no grossly visible papillary tumors within 90 days prior to registration.
* Patients with T1 disease must have cross-sectional imaging of abdomen/pelvis demonstrating no evidence of nodal involvement or metastatic disease (MRI or CT scan) within 90 days prior to registration. Patients with T1 disease must have re-resection confirming ≤ T1 disease within 90 days prior to registration.
* Patients must no have received prior intravesical BCG

Exclusion Criteria:

* Have muscle-invasive or higher (≥T2) bladder cancer
* Unable to give informed consent
* Age 17 or younger
* Taking oral glucocorticoids at the time of registration
* Another cancer requiring active treatment (except basal cell carcinoma or squamous cell carcinoma of the skin)
* Patients at risk of pregnancy that are unwilling or unable to take effective contraception during the study period, or patients that are nursing during the study period. Women/ Men of reproductive potential must have agreed to use an effective contraceptive method or will be considered ineligible for study participation.
* Evidence of nodal involvement or metastatic disease (MRI or CT scan) within 90 days prior to registration
* History of prior intravesical BCG
* History of prior Rapamycin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Determine 1-year Recurrence Free Survival (RFS) rate | 1 year
  The primary analysis will be the estimation of the RFS rate with the 95% confidence interval and comparison of the rate to the historical rate of 68% using the single arm log-rank test (one-sided alpha = 0.05). If the observed rate of RFS is 80% the expected number of events is about 20-28. Recurrence confirmed by pathologic examination of biopsied tissue.
Change in Urinary Quality of Life | Scored at baseline and months 3, 6, 12 and 24. For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  Urinary Quality of Life measured using the urinary domain of the QLQ-BLS24 Index (a 24-item questionnaire that measures quality of life as it relates to urinary symptoms, sexual function, and bother domains). QLQ-BLS24 with a scale ranging from 24-96, and higher scores are worse.
Change in Cognitive Function | EXIT will be scored at baseline and on months 12 and 24.For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  Cognitive function will be measured throughout the study period using EXIT. The EXIT is a brief 25-item interview that will be used by trained research staff to evaluate executive cognitive dysfunction of subjects.
Change in Cognitive Function | SLUMS will be scored at baseline and on months 12 and 24.For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  Cognitive function will be measured throughout the study period using St. Louis University Mental Status exam (SLUMS). The SLUMS exam will be used to evaluate memory, digit span and animal fluency.
Change in Cognitive Function | TAPS will be scored at baseline and on months 6, 12, and 24. For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  Cognitive function will be measured throughout the study period using Texas Assessment of Processing Speed (TAPS). The TAPS test will evaluate digit/symbol coding.
Change in cytoscopy consistent with recurrence (time to recurrence) | Patients will undergo office-based cystoscopy with urine cytology every 3 months for the first 2 years, then every 6 months for 2 years, and at year 5, with biopsies per standard of care if necessary.
  Change in cytoscopy results from baseline consistent with recurrence, confirmed by pathologic examination of biopsied tissue.
Change in Short Physical Performance Battery | SPPB will be scored at baseline and on months 6, 12, and 24. For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  The Short Physical Performance Battery (SPPB) consists of a balance test looking at the ability to maintain three standing positions for 10 seconds, a timed 4-meter walk in which subjects perform their walk at their preferred walking speed, and a chair stand test that times the ability of the subject to arise from a chair 5 times without using their arms. Each section is scored out of 4 points, for a total possible score of 12 points. This test provides information on several motor domains such as static and dynamic balance, coordination, and strength of lower limbs. Lower scores may be associated with increased disability risk. The SPPB and Handgrip Strength are physical assessments.
Change in Handgrip Strength | Handgrip Strength will be scored at baseline and on months 6, 12, and 24. For any subject who has a recurrence after enrollment, but prior to completing a full year of dosing at Visit 6, this will also be measured at the End of Treatment visit.
  When measuring handgrip strength, the subject will be seated in a chair with the forearm at a 90-degree elbow bend. Three consecutive grip strengths will be completed with a standard grip strength dynamometer for both hands. The Handgrip Strength and SPPB are physical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Svatek, MD, MSC, Principal Investigator — UT Health San Antonio
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health San Antonio, San Antonio, Texas